CLINICAL TRIAL: NCT02321111
Title: The Role of TLR4 on Lipid-Induced Insulin Resistance
Acronym: Eritoran1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC20140497H
Record Dates: First submitted 2014-10-29; First posted 2014-12-22 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Insulin Sensitivity
Keywords: Insulin signaling and glucose disposal in muscle; Hepatic insulin sensitivity; TLR4 signaling and inflammatory gene expression; Plasma cytokine concentration; Intramyocellular diacylglycerol and ceramide content
MeSH Terms: conditions — Insulin Resistance | interventions — eritoran; E5564; Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- D5W (5% Dextrose in water) + Saline (Active Comparator): IV administration of 5% Dextrose in water/D5W (vehicle) 12 mg every 12 hours plus Saline infusion at a rate of 30 mL/hour
  Interventions: Drug: D5W (5% Dextrose in water)
- D5W (5% Dextrose in water) + Intralipid (Active Comparator): IV Administration of 5% Dextrose in water /D5W (vehicle) 12 mg plus Intralipid infusion at a rate of 30 ml/hour
  Interventions: Drug: D5W (5% Dextrose in water)
- Eritoran + Intralipid (Active Comparator): IV administration of Eritoran 12 mg every 12 hours plus Intralipid infusion at a rate of 30 ml/hour
  Interventions: Drug: Eritoran

INTERVENTIONS:
Drug: Eritoran — Eritoran = E5564 Eritoran is a pharmacologic inhibitor of TLR4.
  Other Names: E5564
  Arms: Eritoran + Intralipid
Drug: D5W (5% Dextrose in water) — D5W = 5% Dextrose Water Vehicle
  Other Names: Vehicle
  Arms: D5W (5% Dextrose in water) + Intralipid; D5W (5% Dextrose in water) + Saline

SUMMARY:
The purpose of this study is to determine whether pharmacologic inhibition of Toll-like receptor 4 (TLR4) with eritoran for injection (E5564) prevents lipid-induced insulin resistance in lean, normal glucose tolerant (NGT) subjects.

DETAILED DESCRIPTION:
E5564 = Eritoran

ELIGIBILITY:
Inclusion Criteria:

* Subjects capable of giving informed consent.
* lean (BMI <26 kg/m2)
* normal glucose-tolerant subjects (completers) without a family history of Type 2 diabetes mellitus (DM)
* Both genders. (50% males)
* Age = 18-65 years. Older subjects are excluded because aging is a pro-inflammatory state.
* All ethnic groups
* Premenopausal women in the follicular phase, non-lactating, and with a negative pregnancy test. Postmenopausal women on stable dose of or not exposed to hormone replacement for >=6 months.
* Lab: Hematocrit >=34%, serum creatinine <=1.4 mg/dL, normal electrolytes, urinalysis, and coagulation tests. Liver function tests up to 2x normal range.
* Stable body weight (+/-1%) for >=3 months.
* One or less sessions of strenuous exercise/wk for last 6 months.

Exclusion Criteria:

* Presence of diabetes or impaired glucose tolerance based on ADA criteria;
* Current treatment with drugs known to affect glucose and lipid homeostasis. Subjects on a stable dose of statin (>3months) are eligible.
* Non-steroidal anti-inflammatory drugs or systemic steroid use for more than 1 week within 3 months.
* Current treatment with anticoagulants (warfarin). Aspirin (up to 325 mg) and clopidogrel will be permitted if these can be held for seven days prior to the biopsies.
* History of heart disease (New York Heart Classification greater than class II; more than non-specific ST-T wave changes on the ECG), peripheral vascular disease, pulmonary disease, smokers.
* Poorly controlled blood pressure (systolic BP>160, diastolic BP>90 mmHg).
* Active inflammatory, autoimmune, infectious, hepatic, gastrointestinal, malignant, and psychiatric disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Musi, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Audie L. Murphy VA Hospital, STVHCS, San Antonio, Texas, United States

REFERENCES:
- [Derived] Liang H, Sathavarodom N, Colmenares C, Gelfond J, Espinoza SE, Ganapathy V, Musi N. Effect of acute TLR4 inhibition on insulin resistance in humans. J Clin Invest. 2022 Nov 1;132(21):e162291. doi: 10.1172/JCI162291. PMID 36066991

RESULTS

PARTICIPANT FLOW:
Groups:
- Eritoran/Lipid Then D5W/Saline Then D5W/Lipid: Subjects randomized to receive Eritoran/Lipid first then D5W/Saline then D5W/Lipid
- D5W/Saline Then D5W/Lipid Then Eritoran/Lipid: Subjects randomized to receive D5W/Saline first then D5W/Lipid then Eritoran/Lipid
- D5W/Lipid Then D5W/Saline Then Eritoran/Lipid: Subjects randomized to receive D5W/Lipid first then D5W/Saline then Eritoran/Lipid
- D5W/Lipid Then Eritoran/Lipid Then D5W/Saline: Subjects randomized to receive first D5W/Lipid then Eritoran/Lipid then D5W/Saline
- Eritoran/Lipid Then D5W/Lipid Then D5W/Saline: Subjects randomized to receive Eritoran/Lipid then D5W/Lipid then D5W/Saline
- D5W/Saline Then Eritoran/Lipid Then D5W/Lipid: Subjects randomized to receive D5W/Saline then Eritoran/Lipid then D5W/Lipid
Period: Infusion1
Arm/Group | Eritoran/Lipid Then D5W/Saline Then D5W/Lipid | D5W/Saline Then D5W/Lipid Then Eritoran/Lipid | D5W/Lipid Then D5W/Saline Then Eritoran/Lipid | D5W/Lipid Then Eritoran/Lipid Then D5W/Saline | Eritoran/Lipid Then D5W/Lipid Then D5W/Saline | D5W/Saline Then Eritoran/Lipid Then D5W/Lipid
Started | 1 | 4 | 4 | 1 | 0 | 0
Completed | 1 | 4 | 4 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout1 (3-4weeks Between Infusions)
Arm/Group | Eritoran/Lipid Then D5W/Saline Then D5W/Lipid | D5W/Saline Then D5W/Lipid Then Eritoran/Lipid | D5W/Lipid Then D5W/Saline Then Eritoran/Lipid | D5W/Lipid Then Eritoran/Lipid Then D5W/Saline | Eritoran/Lipid Then D5W/Lipid Then D5W/Saline | D5W/Saline Then Eritoran/Lipid Then D5W/Lipid
Started | 1 | 4 | 4 | 1 | 0 | 0
Completed | 1 | 4 | 4 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Infusion2
Arm/Group | Eritoran/Lipid Then D5W/Saline Then D5W/Lipid | D5W/Saline Then D5W/Lipid Then Eritoran/Lipid | D5W/Lipid Then D5W/Saline Then Eritoran/Lipid | D5W/Lipid Then Eritoran/Lipid Then D5W/Saline | Eritoran/Lipid Then D5W/Lipid Then D5W/Saline | D5W/Saline Then Eritoran/Lipid Then D5W/Lipid
Started | 1 | 4 | 4 | 1 | 0 | 0
Completed | 1 | 4 | 4 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout2 (3-4weeks Between Infusions)
Arm/Group | Eritoran/Lipid Then D5W/Saline Then D5W/Lipid | D5W/Saline Then D5W/Lipid Then Eritoran/Lipid | D5W/Lipid Then D5W/Saline Then Eritoran/Lipid | D5W/Lipid Then Eritoran/Lipid Then D5W/Saline | Eritoran/Lipid Then D5W/Lipid Then D5W/Saline | D5W/Saline Then Eritoran/Lipid Then D5W/Lipid
Started | 1 | 4 | 4 | 1 | 0 | 0
Completed | 1 | 4 | 4 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Infusion3
Arm/Group | Eritoran/Lipid Then D5W/Saline Then D5W/Lipid | D5W/Saline Then D5W/Lipid Then Eritoran/Lipid | D5W/Lipid Then D5W/Saline Then Eritoran/Lipid | D5W/Lipid Then Eritoran/Lipid Then D5W/Saline | Eritoran/Lipid Then D5W/Lipid Then D5W/Saline | D5W/Saline Then Eritoran/Lipid Then D5W/Lipid
Started | 1 | 4 | 4 | 1 | 0 | 0
Completed | 1 | 4 | 4 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lean Subjects: Ten lean subjects were randomized to receive 3 infusions in different order.
Arm/Group | Lean Subjects
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.8 (2.2)
HbA1c [Mean (Standard Deviation); unit: Percentage of glycated hemoglobin] | 5.5 (0.3)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] | 5.5 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Eritoran on Muscle Insulin Sensitivity
Description: Muscle insulin sensitivity = muscle insulin sensitivity is determined by euglycemic hyperinsulinemic clamp procedure. M value (mg glucose / kg of body weight / minute) calculated from the clamp is measured. Higher M value indicates better insulin sensitivity. There is no established reference range.
Time Frame: 72 hours
Measure: Mean (Standard Error); unit: mg/kg/min
Arm/Group | D5W (5% Dextrose in Water) + Saline | D5W (5% Dextrose in Water) + Intralipid | Eritoran + Intralipid
Number analyzed (Participants) | 10 | 10 | 10
mg/kg/min | 11.9 (0.6) | 10.2 (0.7) | 9.8 (0.6)
Statistical Analysis 1: Comparison: D5W (5% Dextrose in Water) + Saline vs D5W (5% Dextrose in Water) + Intralipid vs Eritoran + Intralipid; Test type: Other — ANOVA; p = 0.02, ANOVA

2. Primary Outcome: Effect of Eritoran on Hepatic Insulin Sensitivity
Description: Hepatic insulin sensitivity = is determined by euglycemic hyperinsulinemic clamp procedure. Endogenous glucose production or EGP (mg/kg/min) calculated from the clamp is measured. Lower EGP indicates better hepatic insulin sensitivity. There is no established reference range.
Time Frame: 72 hours
Measure: Mean (Standard Error); unit: mg/kg/min
Arm/Group | D5W (5% Dextrose in Water) + Saline | D5W (5% Dextrose in Water) + Intralipid | Eritoran + Intralipid
Number analyzed (Participants) | 10 | 10 | 10
mg/kg/min | 2.2 (0.1) | 2.3 (0.1) | 2.2 (0.0)

3. Secondary Outcome: Effect of Eritoran on TLR4 Expression on Peripheral Blood Monocytes
Description: TLR4 expression on the peripheral blood monocytes is determined by flow cytometry using arbitrary units. Higher TLR4 expression indicates higher inflammatory response. There is no reference range.
Time Frame: 72 hours
Population: Data from 1 subject were not collected due to instrument failure. Therefore, data from 9 subjects were reported.
Measure: Mean (Standard Error); unit: AU
Arm/Group | D5W (5% Dextrose in Water) + Saline | D5W (5% Dextrose in Water) + Intralipid | Eritoran + Intralipid
Number analyzed (Participants) | 9 | 9 | 9
AU | 1.1 (0.1) | 1.2 (0.2) | 1.1 (0.1)

4. Secondary Outcome: Effect of Eritoran on Plasma Cytokine Concentration
Description: TNF-alpha levels (tumor necrosis factor-alpha) are determined by ELISA. Higher level indicates higher inflammatory response. There is no established reference range.
Time Frame: 72 hours
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | D5W (5% Dextrose in Water) + Saline | D5W (5% Dextrose in Water) + Intralipid | Eritoran + Intralipid
Number analyzed (Participants) | 9 | 9 | 9
pg/ml | 1.6 (0.2) | 2.0 (0.3) | 2.0 (0.1)

5. Secondary Outcome: Effect of Eritoran on Intramyocellular Diacylglycerol and Ceramide Content
Description: Intramyocellular diacylglycerol and ceramide content are determined by mass spectrometry. Higher levels have been associated with diabetes.
Time Frame: 72 hours
Population: Data were not collected due to lack of funding.
Arm/Group | D5W (5% Dextrose in Water) + Saline | D5W (5% Dextrose in Water) + Intralipid | Eritoran + Intralipid
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to 20 months
Arm/Group | D5W (5% Dextrose in Water) + Saline | D5W (5% Dextrose in Water) + Intralipid | Eritoran + Intralipid
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 7/10 | 10/10 | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | D5W (5% Dextrose in Water) + Saline (N=10) | D5W (5% Dextrose in Water) + Intralipid (N=10) | Eritoran + Intralipid (N=10)
Phlebitis Grade 1, 2, or 3 (Vascular disorders) | 6 | 8 | 10
Bruising (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypokalemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Dizziness (Nervous system disorders) | 0 | 1 | 1
Upper respiratory illness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT02321111/Prot_SAP_000.pdf